CLINICAL TRIAL: NCT04772599
Title: Measurement of Noradrenaline Concentrations Using Different Dilution Methods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7632
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Arterial Hypertension
Keywords: Noradrenaline; Norepinephrine; Concentration of noradrenaline; Vasopressor; Baby-noradrenaline; Dilution of Noradrenaline
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Norepinephrine is the vasopressor of choice for the treatment of peri-anesthetic arterial hypotension. The use of this drug at significantly lower concentrations (dilution factor between 40 and 200) than the commercial preparation is increasingly common in the operating room ("baby-noradrenaline").

In addition, dilution errors are potentially serious for the patient (hypertensive peak) The preparation of precise dilutions is an important factor for the safe use of this medically In this study, the investigators wish to compare the dilution method of the protocol with another method of preparation (left to the free choice of the participant).

ELIGIBILITY:
Inclusion criteria:

* Adult person,
* Employee of Strasbourg University Hospitals,
* Likely to have to prepare anesthesia drugs in the operating room (intern, hospital student, IADE, IADE student)

Exclusion criteria:

- Subject's refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Employee of the University Hospitals of Strasbourg accepting to participate in the study
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of noradrenaline concentrations using different dilution methods | 1 hour after the preparation of the noradrenaline solutions
  Measurement methods:
  * High performance liquid chromatography
  * Measurement of the concentration of noradrenaline in the biochemical laboratory of the University Hospitals of Strasbourg

CONTACTS AND LOCATIONS:
Locations (1):
- Strasbourg University Hospitals - Anesthesia-intensive care unit, Strasbourg, France